CLINICAL TRIAL: NCT00674336
Title: Norwalk Virus Inactivation by High Hydrostatic Pressure Processing: A Comprehensive and Integrated Program for Research and Outreach
Brief Title: Infectivity of Norovirus in Shellfish Treated With High Hydrostatic Pressure Processing-Human Challenge Study
Acronym: Shellfish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Christine Moe, PhD, Gangarosa Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 0551-2006; RSPHGH-CLM-2007-NoVSHELLFISH (Other: Other)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Norovirus; Gastroenteritis; Clinical Trial; Stomach flu; Oysters; Shellfish; high hydrostatic pressures
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shellfish with Norovirus (Experimental): We dosed shellfish with Norovirus and challenged human volunteers with Shellfish that had norovirus
  Interventions: Procedure: High Hydrostatic Pressure Processing

INTERVENTIONS:
Procedure: High Hydrostatic Pressure Processing — High Hydrostatic Pressure Processing is a technology, used in the food service industry, where foods are subjected to high pressure. These high pressures kill many pathogens without affecting the quality of the food.
  Other Names: HPP

SUMMARY:
Norwalk virus and related "Norwalk-like viruses" are the most common cause of outbreaks of stomach sickness (nausea, vomiting, diarrhea) in older children and adults in the United States. These viruses are sometimes found in drinking water, ice, shellfish and in other foods. They can be spread easily from contact with water, food, objects or hands that have even small amounts of feces from someone who was sick.

The purpose of this research study is to the effectiveness of high hydrostatic pressures processing (HPP) treatment on norovirus infected shellfish. Norwalk virus can survive in shellfish and still be able to cause sickness. HPP inactivates microorganisms living both on the surface and on the interior of the food. The goal of the study is to determine whether HPP treatment on oysters spiked with norovirus will reduce infection rates in people consuming raw infected oysters.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer
* Age must be between 18 and 50 years of age

Exclusion Criteria:

* Have a job in which you handle food
* Are a health care worker with direct patient contact
* Work in a child care, elderly care center or if you live with young children or anyone who has a weak immune system
* Are not willing or able to wash your hands every time after you go to the bathroom, or before and after you prepare or handle food throughout the whole study
* Are anemic
* Are not willing to give us permission to store and use your data and samples

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Infection with norovirus | Throughout participation in study

CONTACTS AND LOCATIONS:
Overall Officials: Christine Moe, PhD, Principal Investigator — Emory University; George M Lyon III, MD, MMSc, Principal Investigator — Emory University
Locations (1):
- Emory University General Clinical Research Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Leon JS, Kingsley DH, Montes JS, Richards GP, Lyon GM, Abdulhafid GM, Seitz SR, Fernandez ML, Teunis PF, Flick GJ, Moe CL. Randomized, double-blinded clinical trial for human norovirus inactivation in oysters by high hydrostatic pressure processing. Appl Environ Microbiol. 2011 Aug;77(15):5476-82. doi: 10.1128/AEM.02801-10. Epub 2011 Jun 24. PMID 21705552
- [Derived] Williams AM, Ladva CN, Leon JS, Lopman BA, Tangpricha V, Whitehead RD, Armitage AE, Wray K, Morovat A, Pasricha SR, Thurnham D, Tanumihardjo SA, Shahab-Ferdows S, Allen L, Flores-Ayala RC, Suchdev PS. Changes in micronutrient and inflammation serum biomarker concentrations after a norovirus human challenge. Am J Clin Nutr. 2019 Dec 1;110(6):1456-1464. doi: 10.1093/ajcn/nqz201. PMID 31504095